CLINICAL TRIAL: NCT06878170
Title: A First in Human Study to Evaluate the Safety and Immunogenicity of RBM-001 in Healthy Adult Volunteers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rock BioMedical, Inc. (Industry)
Responsible Party: Principal Investigator, Sandra Pagnussat, M.D., Medical Director, QPS Holdings LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4587C240015
Record Dates: First submitted 2025-03-04; First posted 2025-03-14 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Placebo control, double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- RBM-001 Cohort 1 (Active Comparator): Low-dose study vaccine administered via intra-muscular injection.
  Interventions: Biological: RBM-001
- RBM-001 Cohort 2 (Active Comparator): High-dose study vaccine administered via intra-muscular injection.
  Interventions: Biological: RBM-001

INTERVENTIONS:
Biological: RBM-001 — To evaluate the safety and tolerability of the RBM-001 vaccination in healthy adults.

SUMMARY:
A First in Human Study to Evaluate the Safety and Immunogenicity of RBM-001 in Healthy Adult Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female, aged 18 to 55 years old (inclusive) at the Screening visit.
2. Body mass index (BMI) of 18.0 to 32.0 kg/m2 (inclusive) at the Screening visit.
3. Physically and mentally capable of participating in the study and willing to adhere to study procedures.
4. Able to provide signed informed consent.
5. In generally good health with no clinically significant abnormal findings in medical history, physical examination, vital signs, ECG, and clinical laboratory findings at the Screening visit based on the Investigator's judgment.
6. Negative serology test for human immunodeficiency virus (HIV) antigen and antibody, hepatitis B surface antigen, and hepatitis C antibody at the Screening visit.
7. All female subjects must have a negative result of pregnancy test at the Screening visit.
8. Female subject with childbearing potential must be willing to implement adequate, highly effective contraceptive measures from the Screening Visit (unless otherwise stated) through end of study (EOS). Effective birth control includes:

   1. Progesterone implant (in place for at least 3 months prior to the Screening Visit) with condom
   2. Progesterone only hormonal contraception (oral or injectable; used consecutively for at least 3 months prior to the Screening Visit) with condom
   3. Progesterone releasing intrauterine device (IUD; in place for at least 3 months prior to the Screening Visit) with condom
   4. Non-hormonal IUD (in place for at least 3 months prior to the Screening Visit)
   5. Bilateral occlusion/tubal ligation
   6. Azoospermic partner
   7. Combined contraceptives (oral, intravaginal, transdermal, implantable, or injectable; in place for at least 3 months prior to the Screening Visit) plus condom; or
   8. Sexual abstinence as the preferred lifestyle (refraining from heterosexual activity) Women of childbearing potential are those who have not been surgically sterilized (hysterectomy, bilateral salpingectomy and bilateral oophorectomy) or are not postmenopausal, defined as no menses for ≥ 12 months without alternative cause with confirmatory laboratory levels.
9. Male subject who agrees to use an adequate method of contraception during the study period (e.g. barrier contraceptives [male condom]).

Exclusion Criteria:

1. Any medical or psychiatric condition that, in the opinion of the Investigator, may interfere with optimal participation in the study or place the subject at increased risk of Adverse Events (AEs).
2. Suspected or known hypersensitivity (including allergy) to any of the ingredients or components in the study vaccine.
3. History of hypersensitivity or allergy to any vaccine.
4. Current, confirmed or suspected acute COVID-19 with positive test for SARS-CoV-2 virus at the Screening visit or at check-in for each period. Acute infection will be confirmed/excluded via symptoms and COVID-19 PCR or antigen testing, including positive COVID-19 PCR or rapid antigen test result within 3 months prior to Screening, reported verbally.
5. Prior history of heart diseases of concern: history of myocarditis, pericarditis, cardiomyopathy, coronary artery disease (including history of myocardial infarction, unstable angina), Class III and above heart failure, or significant arrhythmias.
6. Medical conditions as a contraindication to the IM vaccination and blood draws, e.g. coagulation disorder.
7. Any abnormality or permanent body art (e.g. tattoo) that would interfere with the observation of local reactions at the injection site (deltoid region).
8. Acute or chronic, clinically significant cardiovascular, pulmonary, hepatic or renal diseases and/or insufficiency as determined by physical examination or laboratory tests.
9. Known or suspected impairment of immunological function, e.g. asplenia/splenectomy or history of autoimmune/immune-mediated diseases or lymphoproliferative disorders.
10. History of any chronic or progressive disease that, according to judgment of the Investigator, could interfere with the study outcomes or pose a threat to the subject's health.
11. History of cancer (except localized skin cancer without metastases) within 5 years prior to the Screening visit.
12. History or presence of heavy smoking (defined as > 10 cigarettes per day; approximately half pack per day) as documented in medical chart or by verbal confirmation at the Screening visit.
13. Documented history of substance or alcohol abuse in the medical chart or by verbal confirmation within 6 months prior to the Screening visit.
14. Corrected QT using Fredericia's formula (QTcF) prolongation > 450 milliseconds in males and >470 milliseconds in females at Screening visit.
15. Abnormal troponin (cardiac troponin; cTN) value at Screening visit.
16. Received any investigational or licensed COVID-19 vaccines within 6 months prior to the Screening visit.
17. Received marketed inactivated vaccines against seasonal influenza within 7 days prior to the study vaccination, any other inactivated vaccination within 14 days prior to the study vaccination, or live or bacterial vaccination within 28 days prior to the study vaccination or plans to receive vaccination during the study period or within the 14 days following study vaccination.
18. Received major surgery or radiation therapy within 3 months prior to the Screening visit.
19. Onset of influenza-like illness as defined by: fever (temperature ≥ 38℃), dry cough, headache, fatigue, respiratory sputum production, dysgeusia, anosmia, shortness of breath, muscle and joint pain, or sore throat within 1 week prior to the Screening visit and within 48-hours of each vaccination. Subject can be re-evaluated after resolution of symptoms within the screening window.
20. Female subject who is pregnant at the Screening visit or planning to be pregnant during the study period.
21. Female subject who is breastfeeding at the Screening visit or plans to breastfeed from the time of the first vaccination through 60 days after the last vaccination.
22. Received any investigational mRNA COVID-19 vaccination within 6 months prior to the Screening visit or have received any other investigational drug or device or have participated in a clinical study within 28 days or 5 half-lives of investigational drug prior to the Screening visit.
23. Any confirmed or suspected abnormal immune function, immunosuppression, or immunodeficiency or received any immunosuppressants (including systemic corticosteroids) or immunomodulators within 3 months prior to the Screening visit.
24. Had donated blood within 2 weeks prior to the Screening visit.
25. Received any blood products or immunoglobulin within 3 months prior to the Screening visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence, severity, and relationship of solicited local and general adverse events (AEs) during the 7 days following each vaccination. | Day 1 to Day 8 after first vaccination, Day 22 to Day 29 after second vaccination
Occurrence, severity, and relationship of unsolicited AEs during the 21 days following each vaccination | Day 1 (post-vaccination) to Day 21 for first vaccination, Day 22 (post-vaccination) to Day 43
Occurrence, severity and relationship of adverse events of special interest (AESIs) from the first vaccination through the 28 days following the second vaccination. | Day 1 through Day 50
Occurrence, severity, and relationship of medically-attended AEs (MAAEs), new-onset chronic medical conditions (NOCMCs), and serious adverse events (SAEs) through the study completion | Day 1 through Day 383 (End of study follow-up period)
Occurrence of clinically significant changes in clinical laboratory results, vital signs results, 12-lead ECG results, and physical examination findings | Day 1 through Day 383 (End of Study)

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of antigen specific antibody | Day -1, Day 8, Day 15, Day 21, Day 29, Day 36, Day 43 and Day 113
The geometric mean fold rise (GMFR) in antigen specific antibody titer from baseline | Day -1, Day 8, Day 15, Day 21, Day 29, Day 36, Day 43 and Day 113
Activation of SARS-CoV-2 specific cytotoxic T-cells and helper T-cells | Day -1, Day 21, Day 43 and Day 113
Assessment of specific cytokine levels from baseline through scheduled timepoints throughout study | Day -1, Day 8, Day 15, Day 21, Day 29, Day 36, Day 43 and Day 113

CONTACTS AND LOCATIONS:
Locations (1):
- QPS Miami, Miami, Florida, United States